# Study Title: The Immune Directed Individualized Elimination Therapy (iDIET) Study

NCT number NCT05543512 Document Date 05/22/2025

# University of North Carolina at Chapel Hill Consent to Participate in a Research Study Adult Participants

Consent Form Version Date: 30Apr2025

IRB Study # 22-0500

Title of Study: An allergen-specific immune signature-directed diet vs sham diet for treatment

of eosinophilic esophagitis: A pilot-feasibility study (iDIET)

Principal Investigator: Evan Dellon

Principal Investigator Department: Medicine-Gastroenterology

Principal Investigator Phone number: (919) 966-2511

Principal Investigator Email Address: evan dellon@med.unc.edu

Funding Source and/or Sponsor: NIH National Institute of Diabetes, Digestive, and Kidney

Diseases (NIDDKD)

Study Contact Telephone Number: (919) 966-8559 Study Contact Email: Lucas plott@med.unc.edu

#### CONCISE SUMMARY

The purpose of this research study is to determine the effectiveness of an allergen-specific immune-signature directed diet in the treatment of patients with Eosinophilic Esophagitis (EoE). Participants will provide blood and biopsies (small tissue samples) for the research study during a clinically scheduled upper endoscopy. The samples will be analyzed by a lab to determine potential food allergens. Participants will be randomized (by chance) to receive a custom diet intervention that requires they exclude their food triggers based on the lab results (if in the active group) or a "sham" diet in which they are provided with a diet that randomly excludes foods without considering their results from the lab. Participants will meet with a dietician to discuss their assigned diet before starting their diet and at 4 and 8 weeks after starting their diet, to check to make sure they are sticking with the diet. Participants will follow their assigned diet for 8 weeks, complete questionnaires, and a food diary. At 8 weeks, participants will return for a follow-up endoscopy as part of their routine clinical care, during which time they will be asked again to provide blood and biopsies for this research study. Participants will have up to 3 inperson visits during the study, and each visit will last up to 1 hour. Participation in the study will last up to 19 weeks, but data will also be collected from participant medical records until the study is closed and will be stored indefinitely and may be shared with other researchers.

Risks of this study are related to blood draw (small risk of fainting or bruising and a 1/1000 risk of infection at the site where the blood is drawn) and biopsies (a very small risk (less than 1%) of perforation (making a tear in the esophagus) or significant bleeding that would require a blood transfusion or other measures to stop the bleeding).

If you are interested in learning more about this study, then please continue to read below.

## What are some general things you should know about research studies?

You are being asked to take part in a research study. To join the study is voluntary.

You may choose not to participate, or you may withdraw your consent to be in the study, for any reason, without penalty.

Research studies are designed to obtain new knowledge. This new information may help people in the future. You may not receive any direct benefit from being in the research study. There also may be risks to being in research studies. Deciding not to be in the study or leaving the study before it is done will not affect your relationship with the researcher, your health care provider, or the University of North Carolina-Chapel Hill. If you are a patient with an illness, you do not have to be in the research study in order to receive health care.

Details about this study are discussed below. It is important that you understand this information so that you can make an informed choice about being in this research study.

You will be given a copy of this consent form. You should ask the researchers named above, or staff members who may assist them, any questions you have about this study at any time.

## What is the purpose of this study?

The purpose of this research study is to determine the effectiveness of an allergen-specific immune-signature directed diet in the treatment of patients with Eosinophilic Esophagitis (EoE). EoE is a disease where the lining of the esophagus (food pipe) becomes swollen and inflamed. The lining contains cells, called eosinophils, which would not normally be there. It is believed this disease is caused by an allergic reaction to something that is eaten or breathed in. EoE can cause trouble swallowing, feeding problems, heartburn, chest pain, or other symptoms.

Diet elimination therapy is one common way to treat the symptoms of EoE by taking certain food groups out of a diet and having an upper endoscopy to see if the esophagus has improved. This therapy can be expensive and take a lot of time, and the usual type of "allergy tests" that are done (for example, the skin prick panel on the arm or the back to see what foods react) are not accurate for finding food allergies in EoE. This is why we are studying this new way to check for EoE-related food allergy triggers. The new method we are studying to identify food triggers involves analyzing your samples in a lab. The methods we are using in the lab are considered a device, and the device is investigational and has not been approved by the FDA.

You are being asked to be in the study because you are between 16 and 80 years old, have a diagnosis of EoE, and are planning to undergo dietary elimination therapy as part of your routine clinical care.

## Are there any reasons you should not be in this study?

You should not be in this study if you:

- 1) Have been treated unsuccessfully with a six-food elimination diet
- 2) Have not been on a stable diet within 4 weeks of your baseline endoscopy for the study, or will be unable to maintain a stable diet for the duration of the study

- 3) Have eosinophilic gastroenteritis
- 4) Have used systemic corticosteroids within 4 weeks of your baseline endoscopy for this study
- 5) Have had an esophageal resection (part of your esophagus removed)
- 6) History of bleeding disorder or esophageal varices
- 7) Current use of blood thinners such as coumadin, warfarin, heparin, and/or novel anticoagulant agents (requires discontinuation of medication within an appropriate time frame for that specific agent and in accordance with standard clinical practice)
- 8) Have medical instability that precludes safely performing an upper endoscopy
- 9) Are unable to read or understand English
- 10) Are pregnant or breastfeeding
- 11) Have a body mass index of less than 17

# How many people will take part in this study?

Approximately 100 people at this institution will take part in this study.

# How long will your part in this study last?

Your participation in this study will last up to 19 weeks depending on turnaround time of lab samples and scheduling of your 8-week follow-up endoscopy for routine clinical care. In addition, upon completing the 8-week follow-up endoscopy, you will return to your routine clinical care and data may be collected from your medical record and used in this study indefinitely. Samples collected as part of this study will be coded and stored indefinitely for future research and may be shared with other researchers.

## What will happen if you take part in the study?

After signing this consent form, you will complete questionnaires and proceed with your upper endoscopy that has been scheduled as part of your routine clinical care. Prior to your endoscopy, if you are a female with reproductive potential and you did not receive a urine pregnancy test as part of your clinical care, then you will complete a urine pregnancy test as part of this study. You will then provide a blood sample for the study. A blood sample will be collected through the intravenous (IV) line (which is placed as part of your clinical care for the procedure). Every effort will be made to collect blood from the IV line. However, if unable to collect the blood sample from the IV line, the study team will ask if they can perform a blood draw to collect the samples. You may also decide to come in for a study-specific visit to complete the blood draw before your clinical endoscopy.

You will proceed with your clinical upper endoscopy. During the upper endoscopy, biopsies will be taken as part of your clinical care. Slides may be cut from your clinical biopsies and used in the study. In addition to clinical biopsies, up to 8 additional biopsies will be taken from your esophagus for use in this study (research biopsies). Baseline demographic and medical history information will also be collected during the visit.

Your samples will then be sent to a lab to be analyzed for food triggers. You will then be randomized by chance 1:1 (50/50 chance) to either receive a diet in which you eliminate all foods that the lab determined were triggers OR a sham (pretend) diet in which you will be assigned to exclude foods without considering your food trigger results from the lab. Neither

you, your health care providers, nor the PI or study coordinators, will know to which group you have been assigned.

Once you have been randomized and your diet is assigned, then you will have a virtual meeting with a dietician (phone or videoconference) to gather information about your baseline diet, discuss your assigned diet, and answer any questions you may have. For 1 week leading up to your visit with the study dietician you will be asked to complete a daily food diary. During the week of daily food diary completion, you will fill out the diary during two weekdays (at least one of which is a workday if you work) and during one weekend day. The daily food records will be provided to the study dietician for review. After meeting with the study dietician to discuss your assigned diet, you will then follow your assigned diet elimination for 8 weeks.

You will complete weekly questionnaires starting one week from beginning your assigned diet through completion of your week 8 endoscopy. The study team will show you how to complete the questionnaires during your initial endoscopy visit, and each week you can choose to complete them on your own, or with a study team member via phone or videoconference to ensure you are completing them correctly.

4 weeks after starting the assigned diet elimination, you will have a virtual check-in visit with the study dietician (phone or videoconference) to assess how well you are sticking to the diet and answer any questions you might have about the diet. For 1 week leading up to your visit with the study dietician you will be asked to complete a daily food diary. During the week of daily food diary completion, you will fill out the diary during two weekdays (at least one of which is a workday if you work) and during one weekend day. The daily food records will be provided to the study dietician for review

At 8 weeks you will return for an upper endoscopy as part of your routine clinical care. You will also have a virtual check-in visit with the study dietician (phone or videoconference) to assess how well you are sticking to the diet. For 1 week leading up to your week 8 endoscopy, you will be asked to complete a daily food diary. During the week of daily food diary completion, you will fill out the diary during two weekdays (at least one of which is a workday if you work) and during one weekend day. The daily food records will be provided to the study team at the week 8 endoscopy.

During this week 8 endoscopy, if you are a female with reproductive potential and you did not receive a urine pregnancy test as part of your clinical care, then you will complete a urine pregnancy test as part of this study. You will then provide a blood sample for the study, and you will proceed with your upper endoscopy. During the upper endoscopy, biopsies will be taken as part of your clinical care. Slides may be cut from your clinical biopsies and used in the study. In addition to clinical biopsies, up to 8 additional biopsies will be taken from your esophagus for use in this study (research biopsies). You will also be asked to complete additional questionnaires.

You will then return to the clinical care of your provider for continued follow-up and treatment of your EoE which could include food re-introduction to confirm whether the foods that were eliminated flare up the EoE when they are added back.

After 8 weeks your active involvement in the study is complete, but information may continue to be collected from your medical record and used in this study until the study is closed. You may also be asked to join other research studies to continue collecting specimens and data about you and your condition.

# What are the possible benefits from being in this study?

Research is designed to benefit society by gaining new knowledge. The benefits to you from being in this study may be improvement in EoE symptoms, as well as learning if there are certain foods that are triggers for your EoE that would not be detected otherwise.

## What are the possible risks or discomforts involved from being in this study?

First, there is a risk of loss of confidentiality. By participating in this project, you agree to allow the research team to gather and store clinical information about you that pertains to your condition. Every effort will be made by the research staff, however, to prevent loss of confidentiality, by keeping all data and records under lock and key, using password-protected computers, and by eventually only referring to your data by an anonymous code number.

Second, there are risks due to the additional biopsies obtained during upper endoscopy (EGD) procedures. The upper endoscopies in this study are all procedures you will be having as part of your routine clinical care and are not specific to your participation in the study. The additional biopsies are the study-specific component. Therefore, risks related to this study are specific to the additional research biopsies only. All other endoscopy risks are reviewed as part of your clinical care and are not considered risks related to participation in this study. The number of biopsies taken for this study is within the spectrum of routine clinical practice for esophageal diseases and EoE in particular. Nevertheless, there is a very small risk (less than 1%) of perforation (making a tear in the esophagus) or significant bleeding that would require a blood transfusion or other measures to stop the bleeding. To minimize this risk, we will actively monitor for any bleeding during the biopsy portion of the procedure, and if bleeding is heavy, we will perform clinically indicated maneuvers to stop the bleeding, and then stop further biopsy procurement.

Third, there are risks due to the blood draw. There is a small risk of fainting or bruising and a 1/1000 risk of infection at the site where the blood is drawn. To reduce these risks, we will attempt to draw blood from the IV started prior to endoscopy (an IV is required for administration of sedation medications) but if unable to draw blood from the IV line, then a separate blood draw may be performed.

Fourth, there is a risk you will be assigned to the sham diet in which you would continue eating foods that may be triggering your EoE symptoms/instructed to eliminate the wrong foods from your diet. Risks of eliminating the wrong food(s) are that your condition may not get better or may worsen.

There may be uncommon or previously unknown risks. You should report any problems to the researcher.

Pregnancy tests will be done on all females who might be able to get pregnant at the start of the study. If not completed as part of your routine clinical care, then the study will pay for these pregnancy tests.

# If you choose not to be in the study, what other treatment options do you have?

You do not have to be in this research study in order to receive treatment. If you do not wish to participate, then you will still proceed with the upper endoscopy that your doctor has ordered. After the procedure, the study doctor will be available to discuss other treatment options with you. The other procedures or treatments that are available include prescription medications, and diet elimination therapy without study participation.

# What if we learn about new findings or information during the study?

You will be given any new information gained during the course of the study that might affect your willingness to continue your participation.

# How will information about you be protected?

Participants will not be identified in any report or publication about this study. We may use coded limited data and/or specimens from this study in future research without additional consent.

Electronic data will be kept on secure password-protected computers. Paper records will be kept in secure and locked areas with access limited to research personnel. All participants will be assigned a unique code that does not include any personal identifiers. A file linking you to your code will be maintained by the principal investigator.

Although every effort will be made to keep research records private, there may be times when federal or state law requires the disclosure of such records, including personal information. This is very unlikely, but if disclosure is ever required, UNC-Chapel Hill will take steps allowable by law to protect the privacy of personal information. In some cases, your information in this research study could be reviewed by representatives of the University, research sponsors, or government agencies (for example, the FDA) for purposes such as quality control or safety.

A copy of this consent form will go in to your medical record. This will allow the doctors caring for you to know what study medications or tests you may be receiving as a part of the study and know how to take care of you for other health problems or needs during the study.

#### What is a Certificate of Confidentiality?

This research is covered by a Certificate of Confidentiality. With this Certificate, the researchers may not disclose or use information, documents or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings in the United States, for example, if there is a court subpoena, unless you have consented for this use.

The Certificate cannot be used to refuse a request for information from personnel of a federal or state agency that is sponsoring the study for auditing or evaluation purposes or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA).

The Certificate of Confidentiality will not be used to prevent disclosure as required by federal, state, or local law, such as mandatory reporting requirements for child abuse or neglect, disabled adult abuse or neglect, communicable diseases, injuries caused by suspected criminal violence, cancer diagnosis or benign brain or central nervous system tumors or other mandatory reporting requirement under applicable law. The Certificate of Confidentiality will not be used if disclosure is for other scientific research, as allowed by federal regulations protecting research subjects or for any purpose you have consented to in this informed consent document.

You should understand that a Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers may not use the Certificate to withhold that information.

# Will my genetic information be shared?

Your blood and tissue samples contain genes that are made of DNA unique to you. To do more powerful research, it is helpful for researchers to share information they get from studying human samples. They do this by putting it into one or more scientific databases, where it is stored along with information from other studies. Researchers can then study the combined information to learn even more about health and disease. If you agree to take part in this study, some of your genetic and health information might be placed into one or more scientific databases. There are many different kinds of scientific databases; some are maintained by this institution, some are maintained by the federal government, and some are maintained by private companies. For example, the National Institutes of Health (an agency of the federal government) maintains a database called "dbGaP." A researcher who wants to study the information must apply to the database. Different databases may have different ways of reviewing such requests. Researchers with an approved study may be able to see and use your information, along with information from many other people. Your name and other information that could directly identify you (such as address or social security number) will never be placed into a scientific database. However, because your genetic information is unique to you, there is a small chance that someone could trace it back to you. The risk of this happening is very small but may grow in the future as technology advances. Researchers will always have a duty to protect your privacy and to keep your information confidential.

Federal law called the Genetic Information Nondiscrimination Act (GINA) generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. GINA does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. GINA also does not protect you against discrimination based on an already-diagnosed genetic condition or disease.

By signing this informed consent document, you agree that some of the information generated by participating in this study and/or a copy of the consent form may be included in your medical record and that this information may be viewed by other physicians or caregivers who provide healthcare services to you. This will allow the doctors caring for you to know what study medications or tests you may be receiving as a part of the study and know how to take care of

you if you have other health problems or needs during the study. Additionally, the information may be shared with your medical insurance plan if the research services provided are billed to your insurance.

# Will you receive results from research involving your specimens?

Throughout the study, you will continue receiving clinically relevant results from biopsies taken as part of your routine clinical care.

At the completion of the entire study, results from your food triggers as analyzed by the laboratory will be communicated to you. Any other or future research with your specimens is not expected to yield new information that would be meaningful to share with you personally. There are no plans to re-contact you or other subjects with information about other research results.

The use of your samples may result in commercial profit. You will not be compensated for the use of your samples other than what is described in this consent form.

You will be asked to sign a separate form ("HIPAA Authorization") to allow researchers to review your medical records.

# What will happen if you are injured by this research?

All research involves a chance that something bad might happen to you. If you are hurt, become sick, or develop a reaction from something that was done as part of this study, the researcher will help you get medical care, but the University of North Carolina at Chapel Hill has not set aside funds to pay you for any such injuries, illnesses or reactions, or for the related medical care. Any costs for medical expenses will be billed to you or your insurance company. You may be responsible for any co-payments and your insurance may not cover the costs of study related injuries.

If you think you have been injured from taking part in this study, call the Principal Investigator at the phone number provided on this consent form. They will let you know what you should do.

By signing this form, you do not give up your right to seek payment or other rights if you are harmed as a result of being in this study.

# What if you want to stop before your part in the study is complete?

You can withdraw from this study at any time, without penalty. The investigators also have the right to stop your participation at any time. This could be because you have had an unexpected reaction, or have failed to follow instructions, or because the entire study has been stopped.

If you withdraw or are withdrawn from this study all data collected up until the point of withdrawal will be retained, however no additional information will be collected unless you provide additional written permission for further data collection at the time of your withdrawal.

The investigator may withdraw you from the study at any time for the following reasons:

- You become pregnant or begin breastfeeding.
- You are not complying with study procedures or the assigned intervention.

- You experience adverse events or other conditions in which the investigator determines continued participation in the study would not be in your best interest.
- Your disease progresses in such a way that the investigator determines participation in the study is no longer in your best interest.
- You meet an exclusion criterion (either newly developed or previously not recognized) that prevents further participation.

# Will you receive anything for being in this study?

You will be receiving up to \$100 for taking part in this study. You will receive \$50 after completing all screening and baseline assessments and upon randomization into the study, and \$50 after completing the week 8 follow-up endoscopy. Any payment provided for participation in this study may be subject to applicable tax withholding obligations.

Your name, address, and U.S. tax payer identification number (SSN or ITIN) are required to process payments and/or to report taxable income to the IRS. You must complete a W-9 (for U.S. persons) or W-8BEN and the Foreign Vendor Withholding Assessment with supporting documents (for non-resident aliens) in order to receive payment for participation.

U.S. person participants must complete Form W-9 in order to receive payment for participation. If payment by UNC equals or exceeds \$600 per calendar year for U.S. persons, UNC will report the amount to the Internal Revenue Service on Form 1099. Nonresident alien participants must complete Form W-8BEN and the Foreign Vendor Withholding Assessment with supporting documents in order to receive payment for participation. Payments to nonresident alien participants may be subject to tax withholding and are generally reported to the Internal Revenue Service on Form 1042-S. This information will not be linked to any of the study data and will only be used for payment purposes.

If you do not provide your SSN or ITIN, or complete the appropriate documentation noted above, we cannot issue you a payment for participation. However, you may still choose to participate in this study.

## Will it cost you anything to be in this study?

If you enroll in this study, you will have costs which include travel and parking for study-specific visits with the study dietician (if not completed virtually via video) or if a separate visit is required for your blood draw if for some reason it is unable to be collected on the day of your clinical endoscopy. All other study interactions will piggy-back on visits already scheduled as part of your routine clinical care.

All tests, visits or procedures other than what is done specifically for this study will be related to medical care that is part of the usual care for your condition and would be suggested even if you decided not to be in the research study. Here are some examples of standard medical care that may be performed within this study and will be billed to you or your insurance as part of routine care for your condition: upper endoscopy; esophageal biopsies taken as part of your clinical care; pathology examination of clinical care biopsies; blood tests; and medications to treat EoE or other GI conditions. You will not be billed for extra analysis of the blood or tissue samples that we collect during this study.

You may also have costs associated with your assigned diet. Depending on the number and type of foods that are eliminated from your diet, the study dietician may advise you to use dietary supplements or substitute certain foods with more expensive ones. You will not be reimbursed by the study for these costs because they are routinely expected for a food elimination diet regardless of your participation in this study.

## Who is sponsoring this study?

This research is funded by National Institutes of Health (NIH) National Institute of Diabetes, Digestive, and Kidney Diseases (NIDDKD). This means that the research team is being paid by the sponsor for doing the study. The researchers do not, however, have a direct financial interest with the sponsor or in the final results of the study.

# What if you have questions about this study?

You have the right to ask, and have answered, any questions you may have about this research. If you have questions about the study (including payments), complaints, concerns, or if a research-related injury occurs, you should contact the researchers listed on the first page of this form.

A description of this clinical trial will be available on www.clinicaltrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

# What if you have questions about your rights as a research participant?

All research on human volunteers is reviewed by a committee that works to protect your rights and welfare. If you have questions or concerns about your rights as a research subject, or if you would like to obtain information or offer input, you may contact the Institutional Review Board at 919-966-3113 or by email to IRB\_subjects@unc.edu.

# **Unencrypted Communication Consent**

The study team will message you by email or text, however you may say "no" to receiving these messages and still participate in this study. These messages may include appointment reminders, requests to contact the study team, or reminders to complete study activities. The study team will ask you to provide your preferred email address or cell phone number. These messages may be sent by the study team's personal electronic devices. If you respond to the message, your message may be received by a study team member's personal device. This means there is the risk your information could be shared beyond you and the study team.

If you wish to stop receiving unprotected communication from the study team or have lost access to your device or email account, please notify the study team using the study contact information on the first page of this consent form.

#### IRB Study # 22-0500

**Title of Study**: An allergen-specific immune signature-directed diet vs sham diet for treatment of eosinophilic esophagitis: A pilot-feasibility study (iDIET)

Principal Investigator: Evan Dellon

| Participant's Agreement: | |
|---|---|
| I have read the information provided above. I have asked all the qu | estions I have at this time. I |
| voluntarily agree to participate in this research study. | |
| Signature of Research Participant | |
| Date | |
| Date | |
| Printed Name of Research Participant | |
| Signature of Research Team Member Obtaining Consent | |
| Signature of Research Team Member Obtaining Consent | |
| Date | |
| Printed Name of Research Team Member Obtaining Consent | |
| Signature of Witness if applicable; e.g. literacy issues, visually imp | |
| sign, witness/interpreter for non-English speaking participants using | g the short form) |
| Date | |
| Printed Name of Witness | |